CLINICAL TRIAL: NCT06012448
Title: The Immunologic Effects of Dupilumab in the Treatment of Dermal Hypersensitivity Reaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Mio Nakamura, Assistant Professor of Dermatology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00227361
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Dermal Hypersensitivity Reaction
Keywords: Skin rash; Dupilumab; Skin biopsies
MeSH Terms: conditions — Exanthema | interventions — dupilumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dupilumab (Experimental): All patients will receive dupilumab.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Patients will start by getting dupilumab 600 milligram (mg) subcutaneously at week 0, followed by 300 mg every 2 weeks starting at week 2. The last dose will be given at week 24.
  In addition, participants will have visits at the research site for examinations, provide health information, laboratory draws, skin biopsies (at certain time points). Participation in the study will last approximately 28 weeks.
  Other Names: Dupixent

SUMMARY:
This research is studying a drug called dupilumab to learn about its safety and its effect as a treatment for participants with dermal hypersensitivity reaction. This study will help better understand why and how dermal hypersensitivity reaction occurs and how dupilumab might help treat this condition.

DETAILED DESCRIPTION:
Dermal hypersensitivity reaction is a skin rash that can happen as a reaction to a known trigger or it can happen for unknown reasons. Not a lot is known about why the rash occurs and what happens to the immune system to cause this rash. Dupilumab, a biologic drug that is given as an injection under the skin, may treat dermal hypersensitivity reaction. This study tries to better understand dermal hypersensitivity reaction and how the immune system responds to dupilumab.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of chronic idiopathic DHR as defined by presence of clinical and histopathologic features of DHR for at least 6 weeks without an underlying cause or associated trigger
* Moderate-to-severe DHR as defined by greater or equal 5% total body-surface-area (TBSA) involvement and IGA of greater or equal to 3.
* Female subjects of childbearing potential (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agree either to commit to true abstinence throughout the study and for 12 weeks after the last study drug injection, when this is in line with the preferred and usual lifestyle of the subject, or to use an adequate and approved method of contraception throughout the study and for 12 weeks after the last study drug injection.
* Subject willing and able to comply with all of the time commitments and procedural requirements of the clinical study protocol.

Exclusion Criteria:

* Subjects meeting 1 or more of the following criteria at screening or baseline:
* Had an exacerbation of asthma requiring hospitalization in the preceding 12 months.
* Reporting asthma that has not been well-controlled (ie, symptoms occurring on >2 days per week, nighttime awakenings 2 or more times per week, or some interference with normal activities) during the preceding 3 months.
* Subjects with a current medical history of chronic obstructive pulmonary disease and/or chronic bronchitis.
* Cutaneous infection within 1 week before the baseline visit, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics, or antifungals within 2 weeks before the baseline visit.
* Confirmed or suspected COVID-19 infection within 4 weeks before the screening or baseline visit.
* Previous treatment with dupilumab.
* Pregnant women (positive urine pregnancy test result at the screening visit or the baseline visit), breastfeeding women, or women planning a pregnancy during the clinical study.
* History of, current, or suspected lymphoproliferative disease or malignancy of any organ system within the last 5 years, except for basal cell carcinoma, squamous cell carcinoma in situ (Bowen's disease), or carcinomas in situ of the cervix that have been treated and have no evidence of recurrence in the last 12 weeks before the baseline visit.
* History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, i.e., monoclonal antibody) or to lidocaine.
* Known active or latent tuberculosis (TB) infection.
* Known or suspected immunosuppression or unusually frequent, recurrent, severe, or prolonged infections as per investigator judgment.
* History of or current confounding skin condition (i.e., active atopic dermatitis, chronic urticaria, psoriasis, cutaneous T-cell lymphoma [mycosis fungoides or Sezary syndrome], contact dermatitis, chronic actinic dermatitis, dermatitis herpetiformis).
* Planned or expected major surgical procedure during the clinical study.
* Currently participating or participated in any other study of a drug or device, within the past 8 weeks before the screening visit, or is in an exclusion period (if verifiable) from a previous study.
* History of alcohol or substance abuse within 6 months of the screening.
* History of poor wound healing or keloid formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Th2 immune cell population in lesional Dermal hypersensitivity reaction (DHR) skin at week 16 compared to week 0. | Week 0, week 16

SECONDARY OUTCOMES:
Changes in Total Body surface area (TBSA) in patients with DHR treated with dupilumab at week 2 from week 0. | Week 0, week 2
  The TBSA involvement of DHR will be assessed by the investigator or trained designee for each part of the body (the possible highest score for each region is head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and will be reported as a percentage of all major body sections combined.
Changes in Total Body surface area in patients with DHR treated with dupilumab at week 8 from week 0. | Week 0, week 8
  The TBSA involvement of DHR will be assessed by the investigator or trained designee for each part of the body (the possible highest score for each region is head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and will be reported as a percentage of all major body sections combined.
Changes in Total Body surface area in patients with DHR treated with dupilumab at week 16 from week 0. | Week 0, week 16
  The TBSA involvement of DHR will be assessed by the investigator or trained designee for each part of the body (the possible highest score for each region is head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and will be reported as a percentage of all major body sections combined.
Changes in Total Body surface area in patients with DHR treated with dupilumab at week 24 from week 0. | Week 0, week 24
  The TBSA involvement of DHR will be assessed by the investigator or trained designee for each part of the body (the possible highest score for each region is head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and will be reported as a percentage of all major body sections combined.
Changes in Investigator Global Assessment (IGA) in patients with DHR treated with dupilumab at week 2 from week 0. | Week 0, 2 weeks
  The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the investigator or trained designee to evaluate the global severity of Dermal Hypersensitivity Reaction and the clinical response to a treatment. Treatment success is defined as 0 (clear) or 1 (almost clear) and a 2-point improvement from baseline.
Changes in Investigator Global Assessment in patients with DHR treated with dupilumab at week 8 from week 0. | Week 0, 8 weeks
  The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the investigator or trained designee to evaluate the global severity of Dermal Hypersensitivity Reaction and the clinical response to a treatment. Treatment success is defined as 0 (clear) or 1 (almost clear) and a 2-point improvement from baseline.
Changes in Investigator Global Assessment in patients with DHR treated with dupilumab at week 16 from week 0. | Week 0, 16 weeks
  The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the investigator or trained designee to evaluate the global severity of Dermal Hypersensitivity Reaction and the clinical response to a treatment. Treatment success is defined as 0 (clear) or 1 (almost clear) and a 2-point improvement from baseline.
Changes in Investigator Global Assessment in patients with DHR treated with dupilumab at week 24 from week 0. | Week 0, 24weeks
  The IGA is a 5-point scale ranging from 0 (clear) to 4 (severe) used by the investigator or trained designee to evaluate the global severity of Dermal Hypersensitivity Reaction and the clinical response to a treatment. Treatment success is defined as 0 (clear) or 1 (almost clear) and a 2-point improvement from baseline.
Changes in Pruritus Numeric Rating Scale (NRS) for average itch intensity at week 2 from week 0. | Week 0, 2 weeks
  This scale is used to report the intensity of pruritus during the last 24 hours. The Average Pruritus NRS (AP NRS) provides a measure of overall pruritus intensity over a given period and has clinical relevance to both subjects and physicians because peak pruritus may show higher intensity but short duration. Participants will select from a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Changes in Pruritus Numeric Rating Scale (NRS) for average itch intensity at week 8 from week 0. | Week 0, 8 weeks
  This scale is used to report the intensity of pruritus during the last 24 hours. The Average Pruritus NRS (AP NRS) provides a measure of overall pruritus intensity over a given period and has clinical relevance to both subjects and physicians because peak pruritus may show higher intensity but short duration. Participants will select from a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Changes in Pruritus Numeric Rating Scale (NRS) for average itch intensity at week 16 from week 0. | Week 0, 16 weeks
  This scale is used to report the intensity of pruritus during the last 24 hours. The Average Pruritus NRS (AP NRS) provides a measure of overall pruritus intensity over a given period and has clinical relevance to both subjects and physicians because peak pruritus may show higher intensity but short duration. Participants will select from a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Changes in Pruritus Numeric Rating Scale (NRS) for average itch intensity at week 24 from week 0. | Week 0, 24 weeks
  This scale is used to report the intensity of pruritus during the last 24 hours. The Average Pruritus NRS (AP NRS) provides a measure of overall pruritus intensity over a given period and has clinical relevance to both subjects and physicians because peak pruritus may show higher intensity but short duration. Participants will select from a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Changes in Pruritus Numeric Rating Scale (NRS) for maximum itch intensity 2 from week 0. | Week 0, 2 weeks
  This scale is used to report the intensity of pruritus during the last 24 hours. The maximum itch intensity will be noted by the participants by indicating on a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Changes in Pruritus Numeric Rating Scale (NRS) for maximum itch intensity 8 from week 0. | Week 0, 8 weeks
  This scale is used to report the intensity of pruritus during the last 24 hours. The maximum itch intensity will be noted by the participants by indicating on a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Changes in Pruritus Numeric Rating Scale (NRS) for maximum itch intensity 16 from week 0. | Week 0, 16 weeks
  This scale is used to report the intensity of pruritus during the last 24 hours. The maximum itch intensity will be noted by the participants by indicating on a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.
Changes in Pruritus Numeric Rating Scale (NRS) for maximum itch intensity 24 from week 0. | Week 0, 24 weeks
  This scale is used to report the intensity of pruritus during the last 24 hours. The maximum itch intensity will be noted by the participants by indicating on a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable'.

CONTACTS AND LOCATIONS:
Overall Officials: Mio Nakamura, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No